CLINICAL TRIAL: NCT03427463
Title: Comparison of 0.1 and 0.05mg Intrathecal Morphine When Administered With a Multimodal Pain Regimen for Post-cesarean Analgesia
Brief Title: Comparison of 0.1 and 0.05mg Intrathecal Morphine for Post-cesarean Analgesia.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Katherine Hatter, MD, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00072393
Record Dates: First submitted 2018-01-16; First posted 2018-02-09 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cesarean Section

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a randomized controlled single-blinded clinical trial with patients being randomized to receive either 0.1 or 0.05 mg of IT morphine.
Who Masked: Participant
Masking Description: Patients will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- receiving 0.1 mg IT morphine (Active Comparator): Patients will receive the standard of care dose 0.1 mg of intrathecal morphine
  Interventions: Drug: receiving 0.1 mg IT morphine
- recieving 0.05 mg IT morphine (Experimental): Patients will receive 0.05 mg of intrathecal morphine
  Interventions: Drug: recieving 0.05 mg IT morphine

INTERVENTIONS:
Drug: receiving 0.1 mg IT morphine — Patients will receive the standard of care dose 0.1 mg of intrathecal morphine
  Arms: receiving 0.1 mg IT morphine
Drug: recieving 0.05 mg IT morphine — Patients will receive 0.05 mg of intrathecal morphine
  Arms: recieving 0.05 mg IT morphine

SUMMARY:
The purpose of this study is to determine the ideal dose of spinal morphine for use in Cesarean section. Spinal anesthesia (single injection in the lower back to numb patients from the waist down) is commonly used in Cesarean section to provide numbness and pain relief during the surgery, and adding morphine to the spinal anesthetic provides long lasting pain relief for up to 24 hours after surgery. The ideal dose of spinal morphine, when given with other types of pain medications such as nonsteroidal anti-inflammatories and acetaminophen, has not been determined. In addition, spinal morphine can have side effects such as nausea and itching, so using a lower dose of morphine may decrease these side effects while providing the same amount of postoperative pain relief. Study participants will be divided into two groups. Group 1 will receive the standard dose of spinal morphine (0.1mg) while Group 2 will receive a lower dose of spinal morphine (0.05mg). Both groups will receive the standard dose of spinal bupivacaine (numbing medication) and spinal fentanyl (short acting pain medication). The additional pain medications (IV Toradol and oral acetaminophen) will be given to both groups after surgery. Pain control and morphine side effects will be compared between the two groups in order to determine the best dose of spinal morphine for cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* any parturient 18 years of age or older
* undergoing elective cesarean delivery under spinal anesthesia
* able to consent to the study and participate in the follow-up.

Exclusion Criteria:

* any known allergy to morphine
* general anesthesia
* urgent or emergent cases
* any bleeding diathesis or other coagulopathy
* known G6PD deficiency
* any known liver disease
* known alcohol abuse or dependence
* HELLP syndrome
* thrombocytopenia or known platelet dysfunction
* history or active gastrointestinal bleeding
* acute kidney injury or chronic renal insufficiency
* contraindication/refusal to spinal anesthestic
* chronic pain
* chronic narcotic use
* illicit drug use
* allergy to any study related medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion criteria consist of any parturient 18 years of age or older who is undergoing elective cesarean delivery under spinal anesthesia and is able to consent to the study and participate in the follow-up.
Enrollment: 229 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine
Started | 115 | 114
Completed | 101 | 100
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine | Total
Number analyzed (Participants) | 101 | 100 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (5.19) | 31.7 (6.07) | 31.6 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 100 | 201
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 97 | 94 | 191
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 61 | 129
  Black/African American | 24 | 31 | 55
  Other | 9 | 8 | 17
Prior C-Section, yes [Count of Participants; unit: Participants] | 65 | 73 | 138

OUTCOME MEASURES:

1. Primary Outcome: Time to First Narcotic Rescue Dose in the First 24 Hours Post-cesarean Delivery.
Description: This is defined as the number of hours until the first rescue dose of medication was given to participants within the first 24-hours post-op.
Time Frame: 24 hours
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine
Number analyzed (Participants) | 101 | 100
hours | NA [NA to NA] — The median wasn't reached in the 0.1 group, therefore 95% CI is not able to be estimated. | 23.5 [14.5 to 38]

2. Secondary Outcome: Time to First Ambulation After C-section
Description: This outcome evaluated the amount of time reported in hours after c-section the patient first ambulated.
Time Frame: up to 48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine
Number analyzed (Participants) | 101 | 100
hours | 13.6 [0.4 to 72.5] | 13.7 [2.42 to 75.0]

3. Secondary Outcome: Opioid Medication Given During the Participant's Hospital Stay.
Description: This outcome looks at whether or not any opioid medications were given during the participant's hospital stay, reporting the number of subjects who received opioid pain medication during the admission.
Time Frame: From the time of the procedure through discharge, up to 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine
Number analyzed (Participants) | 101 | 100
Participants | 74 | 74

4. Secondary Outcome: Subjective Pain Rating Using Visual Analogue Scales (VAS) Ranging From 0-100.
Description: Subjective pain with ambulation reported by participants using visual analogue scales (VAS) ranging from 0-100 at the 24-hour post-op time point and 48-hour post-op time point. The lower the number, the better the outcome.
Time Frame: 24-hours post operatively and 48-hours post operatively
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine
Number analyzed (Participants) | 101 | 100
units on a scale
  24-hours post-op | 47.9 [43.4 to 52.4] | 49.6 [45.1 to 54.1]
  48-hours post-op | 44.2 [39.7 to 48.8] | 45.9 [41.4 to 50.5]

5. Secondary Outcome: Presence of Opiate Side Effects (Nausea, Vomiting, and Pruritus)
Description: The presence of opiate side effects (nausea, vomiting, and pruritus) was evaluated from 0-24 hours post-op.
Time Frame: 24 hours post operavtively
Measure: Number; unit: participants
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine
Number analyzed (Participants) | 101 | 100
participants
  Any post-op nausea and/or vomiting, or itching, yes | 68 | 62
  Post-Op nausea, yes | 21 | 27
  Post-op vomiting, yes | 11 | 12
  Pruritis, yes | 60 | 58

6. Secondary Outcome: Overall Patient Satisfaction With Pain Control
Description: Patients were asked to mark their satisfaction with pain control using a Visual Analog Scale (VAS) from 0-100. The higher the number, the more satisfied they were with the post-op pain control
Time Frame: 48 hours post-op
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine
Number analyzed (Participants) | 101 | 100
units on a scale | 93.75 [75 to 100] | 94.5 [75 to 100]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from randomization through 48-hours postoperatively.
Arm/Group | Receiving 0.1 mg IT Morphine | Recieving 0.05 mg IT Morphine
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/100
Other Adverse Events (participants affected / at risk) | 68/101 | 62/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Receiving 0.1 mg IT Morphine (N=101) | Recieving 0.05 mg IT Morphine (N=100)
Post-Op Nausea (Gastrointestinal disorders) | 21 (21) | 27 (27)
Post-Op Vomiting (Gastrointestinal disorders) | 11 (11) | 12 (12)
Pruritis (Skin and subcutaneous tissue disorders) | 60 (60) | 58 (58)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT03427463/Prot_SAP_000.pdf